CLINICAL TRIAL: NCT00443469
Title: A Randomized Placebo-controlled Trial on the Use of Repetitive Spinal Magnetic Stimulation as a Therapeutic Option in Patients With Intractable Neuropathic Pain of the Lower Limbs
Brief Title: Spinal Magnetic Stimulation in Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: A/Prof Lo YL, Singapore General Hospital, NNI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #64/2006
Record Dates: First submitted 2007-03-04; First posted 2007-03-06 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Neuropathic Pain
Keywords: magnetic stimulation; neuropathic pain; spinal; lower limb; clinical trial
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic Stimulation (Experimental)
  Interventions: Device: magnetic stimulation
- Magnetic Stimulation with tilted coil (Placebo Comparator): Magnetic Stimulation with tilted coil
  Interventions: Device: Magnetic Stimulation with tilted coil

INTERVENTIONS:
Device: magnetic stimulation — SMS was delivered with a repetitive magnetic stimulator connected to a figure of eight coil capable of delivering a maximum output of 2 Tesla per pulse. The coil measured 90 mm in each wing and was centered over the surface landmark corresponding to the cauda equina region. SMS was performed with the patient lying comfortably in the prone position and a soft pillow supported the lower abdomen. The coil was placed flat over the back with the handle pointing cranially. Each patient on active treatment received 200 trains of 5 pulses delivered at 10 Hz, at an interval of 5 s between each train. As this was a pilot study, each only received 1000 pulses in a single session.
  Arms: Magnetic Stimulation
Device: Magnetic Stimulation with tilted coil — The placebo arm consisted of 'sham' SMS delivered with the coil angled vertically and one of the wing edges in contact with the stimulation point. As this coil type allows maximum magnetic flux at the center of the intersection, we believe minimum or no stimulation was effected at the edge of the coil in contact with the patient. Stimulation parameters and duration were unchanged in this arm.
  Arms: Magnetic Stimulation with tilted coil

SUMMARY:
It involves delivering a train of magnetic pulses, 5 at each time, to the brain. In the present study, we are using the same method to treat severe pain due to nerve conditions. You will be given up to 1000 pulses in total over the spine in the lower back (Spinal Magnetic Stimulation or SMS). Each train will be given in 10-second intervals. You will have SMS on a single day. You will be given SMS pulses at 1 or 10 per second. No stimulation will be given over the head.

You will be assessed before and after the study for up to 1 week. Your usual medical treatment will be continued

DETAILED DESCRIPTION:
You must be aware of that this is a placebo-controlled trial. This means that you may either receive real SMS or sham SMS. The latter involves a harmless process of ineffective stimulation, designed for comparison with real SMS. Whether you receive either form of treatment will be assigned randomly, and there will be a 50% chance of being assigned to either.

ELIGIBILITY:
Inclusion Criteria:

* All with neuropathic lower limb pain

Exclusion Criteria:

* Contraindications to magnetic stimulation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Subjective pain score measurements | 4 days
  NAS score

CONTACTS AND LOCATIONS:
Overall Officials: YL Lo, MD, Principal Investigator — National Neuroscience Institute, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore